CLINICAL TRIAL: NCT00650611
Title: A 27-Week Open-Label Trial To Characterize The Safety And Tolerability Of Orally Administered Ziprasidone In Children And Adolescent Subjects With Bipolar I Disorder (Manic Or Mixed), Schizophrenia Or Schizoaffective Disorder
Brief Title: A Study of the Safety and Tolerability of Oral Ziprasidone in Children and Teens With Psychotic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1281123
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Bipolar Disorder; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Dose Ziprasidone (Active Comparator)
  Interventions: Drug: Ziprasidone
- High-Dose Ziprasidone (Active Comparator)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — Period 1: Initial dose of oral ziprasidone suspension 20 mg twice daily, which was titrated up in 20 mg twice daily increments to a maximum dose of 80 mg twice daily by Day 10.
  Period 2: patients could switch to oral capsules or remain on oral suspension; doses were flexibly titrated to between 10 and 80 mg twice daily based on the individual needs of the patient as determined by the investigator; concomitant antidepressants and/or mood stabilizers were allowed during Period 2 but not Period 1.
  Other Names: Geodon, Zeldox
  Arms: High-Dose Ziprasidone
Drug: Ziprasidone — Period 1: Initial dose of oral ziprasidone suspension 10 mg twice daily, which was titrated up in 10 mg twice daily increments to a maximum dose of 40 mg twice daily by Day 10.
  Period 2: patients could switch to oral capsules or remain on oral suspension; doses were flexibly titrated to between 10 and 80 mg twice daily based on the individual needs of the patient as determined by the investigator; concomitant antidepressants and/or mood stabilizers were allowed during Period 2 but not Period 1.
  Other Names: Geodon, Zeldox
  Arms: Low-Dose Ziprasidone

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of oral ziprasidone in children and teens with psychotic disorders

ELIGIBILITY:
Inclusion Criteria:

* Children and teens with Bipolar I Disorder (manic or mixed), schizophrenia or schizoaffective disorder
* Willingness to discontinue all antipsychotic medications during the study period

Exclusion Criteria:

* Patients who are clinically stable on treatments that are well tolerated
* Substance-induced psychotic disorders

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2003-12; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Adverse events at Baseline, Day 4, and Weeks 1, 2, 3, 4, 8, 12, 18, and 27. | 27 weeks
Electrocardiograms and vital signs at Screening, baseline, Day 4, and Weeks 1, 2, 3, 4, 8, 12, 18, and 27. | 27 weeks
Laboratory data at Screening and Weeks 3, 12, and 27. | 27 weeks

SECONDARY OUTCOMES:
Clinical Global Impressions-Improvement (CGI-I) scale scores on Day 4 and at Weeks 1, 2, and 3. | 3 weeks
Mean change from baseline in Childrens' Global Assessment Scale (CGAS) scores on Day 4 and at Weeks 1, 2, 3, 12, and 27. | 27 weeks
Serum concentrations of ziprasidone and its major metabolites at Weeks 1, 3, 12, and 27. | 27 weeks
Mean change from baseline in Clinical Global Impressions-Severity (CGI-S) scale scores on Day 4 and at Weeks 1, 2, 3, 12, and 27. | 27 weeks
Mean change from baseline in Young Mania Rating Scale (YMRS) scores on Day 4 and at Weeks 1, 2, 3, 12, and 27. | 27 weeks
Mean change from baseline in Brief Psychiatric Rating Scale-Anchored (BPRS-A) scores on Day 4 and at Weeks 1, 2, 3, 12, and 27. | 27 weeks
Mean change from baseline in movement disorder rating scale scores at Weeks 3, 12, and 27. | 27 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Altamonte Springs, Florida
  - Pfizer Investigational Site, Libertyville, Illinois
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Belmont, Massachusetts
  - Pfizer Investigational Site, Brighton, Massachusetts
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Turnersville, New Jersey
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Kirkland, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281123&StudyName=A%20study%20of%20the%20safety%20and%20tolerability%20of%20oral%20ziprasidone%20in%20children%20and%20teens%20with%20psychotic%20disorders